CLINICAL TRIAL: NCT06011980
Title: Life-2023-02 Study on the Efficacy of Growth Inhibitors After Endoscopic Treatment of Acute Esophagogastric Variceal Bleeding
Brief Title: Life-2023-02 Esophagogastric Variceal Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0407
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Acute Esophageal Variceal Hemorrhage
MeSH Terms: interventions — Growth Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants in this group will take growth inhibitors for 5 days after endoscopic treatment.
  Interventions: Drug: Growth Inhibitor
- Group B (No Intervention): Participants in this group will not take growth inhibitor treatment after endoscopic treatment.

INTERVENTIONS:
Drug: Growth Inhibitor — growth inhibitors for 250-500μg/h, ivgtt. for 5 days
  Arms: Group A

SUMMARY:
Study on the efficacy of the growth inhibitors after endoscopic treatment of acute esophagogastric variceal bleeding

DETAILED DESCRIPTION:
Participants with acute esophagogastric variceal bleeding in 5 days and under stable status will be included in this study. All the patients will take CTP test to confirm the blood flow status of the portal vein before endoscopic treatment. After that they will be randomly divided into two groups: A. accept growth inhibitors after the endoscopic treatment for 5 days; B. no growth inhibitor will be applied after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* acute esophagogastric bleeding with hepatic cirhosis;
* stable status (no active bleeding)

Exclusion Criteria:

* endoscopic test limitation;
* previous acute esophagogastric bleeding treatment history;
* ICU;
* pregnant;
* Immunity disabled;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
rebleeding rate after the endoscopic treatment in Group A at 1 month | 1 month after the endoscopic treatment
  record the rebleeding incidence in this group A; (Rate A1= the number of rebleeding participants/the number of all the participants)
rebleeding rate after the endoscopic treatment in Group A at 3 months | 3 months after the endoscopic treatment
  record the rebleeding incidence in this group A; (Rate A2= the number of rebleeding participants/the number of all the participants)
rebleeding rate after the endoscopic treatment in Group A at 6 months | 6 months after the endoscopic treatment
  record the rebleeding incidence in this group A; (Rate A3= the number of rebleeding participants/the number of all the participants)
rebleeding rate after the endoscopic treatment in Group B at 1 month | 1 month after the endoscopic treatment
  record the rebleeding incidence in this group B; (Rate B1= the number of rebleeding participants/the number of all the participants)
rebleeding rate after the endoscopic treatment in Group B at 3 months | 3 months after the endoscopic treatment
  record the rebleeding incidence in this group B; (Rate B2= the number of rebleeding participants/the number of all the participants)
rebleeding rate after the endoscopic treatment in Group B at 6 months | 6 months after the endoscopic treatment
  record the rebleeding incidence in this group B; (Rate B3= the number of rebleeding participants/the number of all the participants)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
on request